CLINICAL TRIAL: NCT02091830
Title: Non-surgical Treatment of Knee Osteoarthritis - a Comparison of Effects in 2200 Patients
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Principal Investigator, Ole Simonsen, MD, DMSc, Northern Orthopaedic Division, Denmark
Other Study IDs: The 07 - 11 cohort
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Physical Therapy Modalities; Cortisone; Bro protein, Drosophila

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-surgical treatment
  Interventions: Drug: Paracetamol and nonsteroidal antiinflammatory drug (NSAID); Other: Physiotherapy; Drug: Cortisone Injection; Other: Others

INTERVENTIONS:
Drug: Paracetamol and nonsteroidal antiinflammatory drug (NSAID)
Other: Physiotherapy
Drug: Cortisone Injection
Other: Others

SUMMARY:
The purpose of this study is to assess whether radiographic osteoarthritis severity (OA; Kellgren-Lawrence scale) is associated with self-reported improvement in pain after non-surgical treatments (physiotherapy, pain killers, injection, other treatments).

The hypothesis is that radiographic OA severity is inversely associated with self-reported improvement.

ELIGIBILITY:
Inclusion Criteria:

* Not eligible for at total knee arthroplasty

Exclusion Criteria:

* Ipsilateral knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2200 patients with knee osteoarthritis not eligible for at total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 2262 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Self-reported improvement | 2-5 years after consulting orthopedic surgeon
  Assessed using the question:
  Has your pain improved? Response categories: pain free; better; unchanged; worse

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rathleff, MSc, Study Chair — Department of Occupational Therapy and Physiotherapy, Aalborg University Hospital, Denmark.; Mikkel M Andersen, MSc, Study Chair — Department of Mathematical Sciences, Aalborg University; Ole Simonsen, MD, DMSc, Principal Investigator — Department of Orthopedic Surgery; Christina A Derosche, BSc, Study Chair — Department of Orthopedic Surgery; Signe B Pedersen, Study Chair — Department of Orthopedic Surgery; Søren T Skou, MSc, Study Chair — Orthopedic Surgery Research Unit + Department of Health Science and Technology, Aalborg University
Locations (1):
- Department of Orthopedic Surgery, Aalborg, Denmark